CLINICAL TRIAL: NCT04835818
Title: Clinical Impact on Point-of-Care Multiplex Polymerase Chain Reaction (PCR) Testing for Critically Ill Adult Patients With Community-acquired Pneumonia
Brief Title: Point-of-Care Multiplex for Adult Patients With Severe Community-acquired Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 201901147RIND
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Community-acquired Pneumonia; Critical Illness
Keywords: Community-acquired Pneumonia; Critical Illness; Point-of-care
MeSH Terms: conditions — Community-Acquired Pneumonia; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reporting (Experimental): check point-of-care Multiplex PCR for pneumonia pathogens and report results to primary care physician
  Interventions: Diagnostic Test: Provide the panel report to the primary care physician
- Usual Care (No Intervention): check point-of-care Multiplex PCR for pneumonia pathogens but do NOT report results to primary care physician. Let primary care physician provide usual standard care

INTERVENTIONS:
Diagnostic Test: Provide the panel report to the primary care physician — Point-of-care Multiplex PCR Respiratory Panel (BIOFIRE FilmArray) and Pneumonia Panel results (BIOFIRE FilmArray)
  Arms: Reporting

SUMMARY:
Clinical Impact on Point-of-Care Multiplex PCR Testing for Critically Ill Adult Patients With Community-acquired Pneumonia - A cluster randomization study in ICU units within one medical center.

DETAILED DESCRIPTION:
Point-of-Care Multiplex PCR Testing could narrow down the pathogens causing severe community-acquired pneumonia(CAP). Our hypothesis is that the result of Point-of-Care Multiplex PCR Testing could help primary physician to reduce antibiotics use.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >20 y/o)
* ICU admission for acute respiratory failure due to community-acquired pneumonia by clinical diagnosis
* Treatment with endotracheal Intubation

Exclusion Criteria:

* Aspiration pneumonia (including witnessed aspiration and chronic bedridden status)
* Nosocomial infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Intravenous antibiotic-free day within 14 days | up to 14 days
  days without intravenous antibiotics within 14 days

SECONDARY OUTCOMES:
ICU stay | up to 21 days
  days of stay in ICU
Antibiotic-free day within 21 days | 21 days
  days without antibiotics within 21 days
Intravenous antibiotic-free day within 21 days | up to 21 days
  days without intravenous antibiotics within 21 days
Ventilator-free day within 28 days | up to 28 days
  days without intravenous antibiotics within 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chung Chuang, MD. PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No